CLINICAL TRIAL: NCT04205734
Title: Methotrexate Polyglutamate Measurements in Patients With Inflammatory Bowel Disease
Status: Suspended | Type: Observational
Why Stopped: COVID Restrictions
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Web, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: IRB-P00028947
Record Dates: First submitted 2019-09-17; First posted 2019-12-19 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: IBD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 5 ml of whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MTX Assessment — Measurement of Methotrexate Polyglutamate levels.

SUMMARY:
There are currently no serum levels to help guide appropriate methotrexate therapy. Data from this study will assess the correlation between dosing and whole blood methotrexate(MTX) polyglutamate measurements in children and adolescents with IBD.

DETAILED DESCRIPTION:
This is a cross-sectional study design. Subjects will be requested to provide one blood sample to be collected during the conduct of their routine clinical care. Data related to the diagnosis and interval assessment of enrolled subjects will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* IBD
* Methotrexate Therapy

Exclusion Criteria:

* Inability to provide relevant samples

Ages: 1 Year to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with IBD being treated with methotrexate (oral or subcutaneous)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Methotrexate Polyglutamate Level | Samples will collected within 16 weeks of consent.
  Measurement of Methotrexate Polyglutamate Levels

SECONDARY OUTCOMES:
The correlation between Methotrexate Polyglutamate Levels and Lab Parameters | Samples will collected within 16 weeks of consent.
  Compare the relationship between Methotrexate Polyglutamage levels and ESR,CRP, Hemoglobin, and Albumin
The correlation between Methotrexate Polyglutamate Levels and Clinical History | Samples will collected within 16 weeks of consent.
  Do Methotrexate Polyglutamate Levels Predict Clinical Outcome as Measured by Disease Activity Indices, including PUCAI for ulcerative colitis and PCDAI for patients with Crohn Disease

CONTACTS AND LOCATIONS:
Overall Officials: PAUL A RUFO, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided